CLINICAL TRIAL: NCT05683704
Title: Phase 2 Multi-center Randomized Study to the Efficacy and Safety of AK105 Combined With Anrotinib Hydrochloride in Patients With Recurrent/Refractory Classical Hodgkin's Lymphoma
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-AK105-II-05
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-04

CONDITIONS: Recurrent/Refractory Classical Hodgkin's Lymphoma
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: AK105，Anrotinib hydrochloride — AK105 administered IV at day 1 every 3 weeks for 8-12 cycles Anrotinib administered PO at day 1-14 every 3 weeks for 8-12 cycles

SUMMARY:
This study is a single arm, open, multi center phase II exploratory study. To evaluate the efficacy and safety of AK105 combined with androtinib hydrochloride capsule in patients with relapsed/refractory classical Hodgkin's lymphoma (relapse or progression after autologous stem cell transplantation, or relapse progression after autologous stem cell transplantation but ≥ 1 line systemic multi drug combination chemotherapy). After screening, the subjects met the inclusion criteria and did not meet the exclusion criteria, and then entered the treatment period. They received AK105 injection (once every three weeks, 200mg/time, intravenous infusion) combined with androtinib hydrochloride capsule (once a day, 10mg each time, and stopped for one week for two consecutive weeks). Every 21 days was a treatment cycle until disease progression/intolerance occurred or the sponsor terminated the study. Patients with complete remission (CR) continue to receive 4 cycles of treatment, and then further consolidate treatment every 9 weeks within 1 year of continuous CR, and can stop treatment after 1 year of continuous CR. At the end of the trial, the subjects who can still benefit from the study treatment as judged by the investigator will continue to be provided with the trial drug. The longest administration time of AK105 combined with androtinib hydrochloride capsules shall not exceed 2 years.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all following criteria to be enrolled in the study:

1. Subjects volunteered to join the study and signed the informed consent form, with good compliance;
2. Age: 18-75 (when signing the informed consent form); ECOG score: 0 or 1; The expected life span is more than 3 months;
3. The patient was diagnosed as classical Hodgkin's lymphoma (cHL) by histopathology (the histopathological diagnosis is based on the pathological specimen of tumor tissue within 3 years before the first administration, and confirmed by the center; if more than 3 years later, the patient needs to be diagnosed by biopsy in the research center);
4. The subject must be a cHL with recurrence (disease progression confirmed after recent treatment) or intractable (complete or partial remission failed after recent treatment), and must meet any of the following criteria: a) receive autologous stem cell transplantation after rescue chemotherapy, and then relapse or progress; b) For subjects who cannot or do not want to receive autologous stem cell transplantation, they are required to have received ≥ first-line standard systemic treatment (including PD-1 treatment); For patients who are difficult to treat, it means that the course of treatment ≥ 2 cycles fails to reach PR, or the treatment ≥ 4 cycles fails to reach CR. If the best effect or the reason for the end of treatment is PD, the number of courses of treatment is not required; For patients with recurrence, they have at least received first-line chemotherapy in the near future before recurrence;
5. Those who have used chemotherapy drugs before the first administration need to stop taking drugs for more than 4 weeks (mitomycin or nitrosoureas, more than 6 weeks), those who have received surgery, molecular targeted therapy, traditional Chinese medicine treatment with anti-tumor indications, and radiotherapy need to stop taking drugs for more than 4 weeks, and those who have used antibody drugs (such as brentuximab vedotin) need to stop taking drugs for more than 12 weeks, In addition, all adverse events (except hair loss) occurred in the treatment have been stabilized and returned to the standard level of admission and discharge or ≤ Grade 1 toxicity (NCI CTCAE Version 5.0);
6. According to CT or MRI evaluation, there is at least one tumor lesion that can be measured by imaging in two vertical directions (according to the 2014 Lugano standard, the length of intranodal lesions is>15mm, and the longest diameter of extranodal lesions is>10mm);
7. The main organs function well and meet the following standards:

   i. The blood routine examination was in line (no blood transfusion and correction with hematopoietic stimulator drugs within 14 days before screening): hemoglobin (HGB) ≥ 80 g/L; Neutrophil absolute value (NEUT) ≥ 1.0 × 109/L； Platelet count (PLT) ≥ 80 × 109/L； ii. Biochemical examination shall meet the following requirements: total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (lymphoma involving liver or biliary obstruction ≤ 5 × ULN）； Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance ≥ 50ml/min; iii. The blood coagulation function test shall meet the following requirements: prothrombin time (PT), activated partial thromboplastin time (APTT), and international normalized ratio (INR) ≤ 1.5 × ULN (without anticoagulation treatment); Iv. Color Doppler echocardiography evaluation: left ventricular ejection fraction (LVEF) ≥ 50%.
8. Female subjects of childbearing age should agree to use contraceptive measures (such as intrauterine device, contraceptive pill or condom) during the study period and within 6 months after the end of the study; The serum or urine pregnancy test was negative within 7 days before the study was included, and must be non lactating subjects; Male subjects should agree to use contraception during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

Presence of any of the following will exclude a patient from enrollment:

1. Nodular lymphoid mainly Hodgkin's lymphoma or gray area lymphoma;
2. Classical hodgkin's lymphoma involves the central nervous system;
3. Participated in experimental drug research or received research treatment within 4 weeks before the first administration, or received anti angiogenesis related drug treatment in the past (including but not limited to bevacizumab, etc.);
4. Subjects with or suspected of active autoimmune diseases, or who have suffered from autoimmune diseases and are at high risk of recurrence, including but not limited to immune related neurological diseases, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain Barre syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma Inflammatory bowel disease includes Crohn's disease and ulcerative colitis, autoimmune hepatitis Toxic epidermal necrolysis (TEN) or Stevens Johnson syndrome, etc. (Note: subjects with vitiligo, eczema, and type I diabetes controlled by hormone replacement therapy and/or physiological corticosteroids can be included in the group. For subjects with rheumatoid arthritis and/or other joint diseases, S-J syndrome, or psoriasis that can be controlled by local medication, or subjects with positive serological tests, such as antinuclear antibody (ANA) Or subjects with positive antithyroid antibody should evaluate whether there is target organ involvement and whether systemic treatment may be required. Exclude subjects with target organ involvement and who need systemic treatment);
5. Subjects who need to use glucocorticoid (>10mg/day equivalent dose of prednisone) or other immunosuppressive drugs for systemic treatment within 14 days before the first administration. The following exceptions are excluded: ① If there is no active autoimmune disease, it is allowed to use inhaled or local corticosteroids and the therapeutic dose of prednisone ≤ 10mg/day; ② Local, intraocular, articular cavity, nasal or inhaled corticosteroids (very low systemic absorption); ③ Glucocorticoid as a preventive drug for hypersensitivity (such as drug before CT examination);
6. Inoculate live vaccine or mRNA vaccine within 4 weeks before the first administration;
7. Have received allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
8. Autologous hematopoietic stem cell transplantation was performed within 3 months before the first administration;
9. Known to have active pulmonary tuberculosis;
10. Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases;
11. Subjects with known history of interstitial pneumonia, non infectious pneumonia or highly suspected interstitial pneumonia; Or subjects who may interfere with the detection or treatment of suspected drug-related pulmonary toxicity;
12. Patients with physical evidence or medical history of bleeding; Within 4 weeks before the first administration, any bleeding event ≥ CTC AE level 3 (such as gastrointestinal bleeding, perforation, etc.) occurred;
13. Complicated diseases and medical history:

    1. He has had or is currently suffering from other malignant tumors within 3 years. The following two conditions can be included in the group: for other malignant tumors treated by single operation, the disease free survival (DFS) of 5 consecutive years has been achieved; Cured cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor [Ta (non invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
    2. There are many factors that affect oral medicine (such as inability to swallow, chronic diarrhea and intestinal obstruction);
    3. Those who have a history of abuse of psychotropic substances and are unable to quit or have mental disorders;
    4. Subjects with any severe and/or uncontrollable disease, including:

       1. Poor blood pressure control (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg);
       2. Patients with ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia (including male QTc ≥ 450ms (male), QTc ≥ 470ms (female)) and ≥ grade 2 congestive heart failure (NYHA classification);
       3. Active or uncontrolled serious infection (≥ CTC AE level 2 infection);
       4. Known liver disease history with clinical significance. Including viral hepatitis. People who are known to be carriers of hepatitis B virus (HBV) must be excluded from active HBV infection, that is, HBV DNA is positive (>2500 copies/mL or>500 IU/mL, and greater than the upper limit of normal value); Known hepatitis C virus infection (HCV) and HCV RNA positive (>1 × 103 copies/mL), or other decompensated liver diseases;
       5. Renal failure requiring hemodialysis or peritoneal dialysis;
       6. Subjects with uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
       7. Poor control of diabetes (FBG>10mmol/L);
       8. Routine urine test indicates that urine protein is ≥++, and 24 hour urine protein quantity is confirmed to be greater than 1.0 g;
14. Within 4 weeks before the start of the study treatment, he has received the treatment of Chinese patent drugs with anti-tumor indications specified in the NMPA approved drug manual (including compound cantharis capsule, Kangai injection, Kanglaite capsule/injection, Aidi injection, Brucea javanica oil injection/capsule, Xiaoaiping tablet/injection, cinobufagin capsule, etc.);
15. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the subject or affect the completion of the study, or subjects who believe that there are other reasons that are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | from May 2022 to May 2024
  To evaluate the efficacy of AK105 combined with androtinib hydrochloride capsule in the treatment of patients with recurrent/refractory classical Hodgkin's lymphoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Insititute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided